CLINICAL TRIAL: NCT01979861
Title: A Prospective, Multicenter, Clinical Trial to Evaluate the Safety and Effectiveness of the AEGEA Vapor System for the Treatment of Excessive Uterine Bleeding
Brief Title: Safety & Effectiveness Study of AEGEA Vapor System to Treat Excessive Uterine Bleeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aegea Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SE-3000
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Menorrhagia
Keywords: Endometrial ablation with vapor
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vapor endometrial ablation (Experimental): endometrial ablation using the AEGEA Vapor System
  Interventions: Device: AEGEA Vapor System(TM)

INTERVENTIONS:
Device: AEGEA Vapor System(TM) — vapor endometrial ablation

SUMMARY:
The purpose of this study is to determine if the AEGEA Vapor System for endometrial ablation is safe and effective for reducing menstrual blood loss in women with excessive uterine bleeding (menorrhagia)

DETAILED DESCRIPTION:
This is a single-arm, multi-center study with three years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female subject from (and including) age 30 to 50 years
* Self-reported history of heavy menstrual bleeding in at least 3 of the last 6 months
* Predictable cyclic menstrual cycles over past 6 months
* Excessive uterine bleeding
* Premenopausal at enrollment
* Normal PAP
* Normal endometrial biopsy
* Willing to use reliable contraception
* Not currently taking hormonal medication
* Agree to use sponsor provided catamenial product (sanitary pads/tampons)

Exclusion Criteria:

* Pregnant
* Desires future childbearing
* Presence of an IUD
* Previous endometrial ablation procedure
* Evidence of STI
* Evidence of PID
* Active infection of genitals, vagina, cervix, uterus or urinary tract
* Active endometritis
* Active bacteremia, sepsis or other active systemic infection
* Gynecologic malignancy
* Endometrial hyperplasia
* Known clotting defects or bleeding disorders
* On anticoagulant therapy
* Hemoglobin <8gm/dl
* Prior uterine surgery
* Currently on medication that could thin myometrial muscle
* Severe dysmenorrhea, secondary to adenomyosis
* Abnormal uterine cavity
* Hydrosalpinx
* Uterine length <6cm or >12cm
* Currently in other clinical trial

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12 months
  Reduction of menstrual blood loss

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint | 12 months
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levie, MD, Principal Investigator — Montefiore Medical Center
Locations (15):
- United States (12):
  - Center for Fertility and Women's Health, New Britain, Connecticut
  - Clinical Associates of Orlando, LLC, Orlando, Florida
  - Visions Clinical Research, Wellington, Florida
  - Rosemark WomenCares Specialists, Idaho Falls, Idaho
  - The Advanced Gynecologic Surgery Institute, Naperville, Illinois
  - Basinksi, LLC, Newburgh, Indiana
  - Minnesota Gynecology & Surgery, Edina, Minnesota
  - Mercy Hospital, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Women's Research and Wellness Center/OB-GYN, Durham, North Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Baylor All Saints, Fort Worth, Texas
- Department of Obstetrics and Gynecology, Hamilton, Ontario, Canada
- Hospital Universitario de la Universidad Autonoma de Nuevo Leon, Monterrey, N.l., Mexico
- Isala Klinieken, Zwolle, Overijissel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leyland N, Harris M. Water Vapor Endometrial Ablation for Heavy Menstrual Bleeding: 36-Month Follow-Up of a Prospective, Multicenter Pivotal Clinical Trial. Int J Womens Health. 2021 Feb 10;13:169-176. doi: 10.2147/IJWH.S279864. eCollection 2021. PMID 33603496